CLINICAL TRIAL: NCT06331403
Title: Open Pilot Trial of a Novel Mind-Body Sexual Well-Being Intervention for Female GI Cancer Survivors
Brief Title: Open Pilot Trial of a Mind-Body Sexual Well-Being Intervention for Female GI Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Lucy Finkelstein-Fox, PhD, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-009
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Anal Cancer; Sexual Dysfunction
Keywords: sexual well-being; women's health; colorectal cancer; anal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Anus Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body Sexual Well-Being Group Intervention (Experimental): Participants in the mind-body sexual well-being group intervention arm will participate in 6 weekly group sessions, delivered via videoconferencing, following enrollment. Group sessions will include content related to mind-body medicine (e.g., relaxation, mindfulness, self-compassion) applied to sexual well-being as well as educational information related to women's sexual well-being in cancer survivorship.
  Before and after completing the group program, participants will also complete brief self-assessment questionnaires to measure topics including satisfaction with sexuality, coping, loneliness, concern about body image, and stigma.
  Interventions: Behavioral: Mind-Body Group Intervention

INTERVENTIONS:
Behavioral: Mind-Body Group Intervention — Weekly virtual group meetings with the study interventionist(s) and up to 9 other female cancer survivors over an approximately 6 week period. The group program includes topics related to coping with physical health changes, managing social factors relevant to sexual well-being, and managing thoughts and feelings related to sexual well-being changes.

SUMMARY:
The primary goal of this protocol is to conduct an open pilot to collect initial quantitative and qualitative feedback on the intervention that the investigators are developing. To do so, the investigators will deliver a newly-developed intervention to up to 2 consecutive groups of female colorectal and anal cancer survivors (n = up to 10 per group, total N = up to 20). Participants will provide feedback regarding intervention acceptability, feasibility, and perceived benefit.

To inform plans for ongoing program refinement, the investigators will elicit specific feedback about study assessment tools, recruitment procedures, and group factors. Given the early-stage, open pilot nature of this protocol, the investigators will not set strict criteria to establish feasibility and acceptability but will rather interpret each of these outcomes holistically. Qualitative feedback collected in post-intervention exit interviews will also support understanding of feasibility and acceptability.

As a secondary aim, the investigators will explore the preliminary effects of the intervention on psychosocial measures of satisfaction with sexuality and impact of functional limitations, coping abilities, acceptance of body image changes, loneliness, and anticipated stigma. As noted above, the investigators will not set specific criteria to establish preliminary efficacy, nor will they consider statistical significance as an indicator of the study's efficacy for these outcomes. Instead, the investigators will consider pre-post intervention effect sizes to consider the need for refinement of study procedures/measurement in a future larger trial.

In future, larger-scale, work, the investigators intend to conduct a larger randomized pilot trial to assess intervention acceptability, feasibility, as well as preliminary efficacy on essential outcomes related to sexual well-being.

DETAILED DESCRIPTION:
This is an open pilot trial to gather initial data regarding feasibility, acceptability, and perceived impact of a 6-session mind-body group intervention that the investigators are developing to enhance sexual well-being among post-treatment female colorectal and anal cancer survivors.

The investigators will enroll up to 10 women per group into up to 2 groups (total N = up to 20). The team will run groups consecutively so that any necessary changes from the first open pilot group may be incorporated and re-examined in the second.

Participants will complete informed consent prior to initiation of study procedures. To inform ongoing intervention refinement, the investigators will ask participants to complete approximately 15-minute survey batteries via REDCap at baseline and after the 6-session program, including assessments of intervention feasibility and acceptability as well as psychosocial outcomes. Participants will also be invited to complete a brief qualitative exit interview with a member of the study team, regarding perceived benefit of the intervention as well as and strengths and weaknesses of program content and delivery format to inform ongoing intervention refinement.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* English-speaking
* Aged 18 or older
* Receive any cancer care at MGH-CC sites (Boston, Waltham, Danvers, Newton Wellesley Hospital)
* Completed initial active treatment (i.e., surgery, radiation, chemotherapy) for colorectal or anal cancer approximately 3 months or more prior to enrollment OR diagnosed longer than 3 months ago if in metastatic cancer treatment.

Exclusion Criteria:

* Active psychiatric or cognitive comorbidity that prohibits the capacity to provide informed consent as determined by the study PI, a licensed psychologist, in collaboration with the patient's medical team
* Adults unable to complete study procedures in English.
* Participated in an earlier phase of the research study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Finkelstein-Fox, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: lfinkelsteinfox@mgh.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team
URL: http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Mind-Body Sexual Well-Being Group Intervention: Participants in the mind-body sexual well-being group intervention arm will participate in 6 weekly group sessions, delivered via videoconferencing, following enrollment. Group sessions will include content related to mind-body medicine (e.g., relaxation, mindfulness, self-compassion) applied to sexual well-being as well as educational information related to women's sexual well-being in cancer survivorship.
  Before and after completing the group program, participants will also complete brief self-assessment questionnaires to measure topics including satisfaction with sexuality, coping, loneliness, concern about body image, and stigma.
  Mind-Body Group Intervention: Weekly virtual group meetings with the study interventionist(s) and up to 9 other female cancer survivors over an approximately 6 week period. The group program includes topics related to coping with physical health changes, managing social factors relevant to sexual well-being, and managing thoughts and feelings related to sexual well-being changes.
Period: Overall Study
Arm/Group | Mind-Body Sexual Well-Being Group Intervention
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mind-Body Sexual Well-Being Group Intervention
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 55 [50 to 73]
Sex/Gender, Customized [Number; unit: participants]
  Female gender | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: The primary feasibility metric will be program engagement, quantified as participant rates of intervention attendance (% attending at least 4 of 6 sessions). Given the preliminary, open pilot nature of this protocol, the investigators will not set a priori criteria to establish feasibility but will rather use these data to inform ongoing protocol refinement.
Time Frame: Approximately 6 weeks after the final 6-week (up to N=2 groups) group program begins
Measure: Count of Participants; unit: Participants
Arm/Group | Mind-Body Sexual Well-Being Group Intervention
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Acceptability of Intervention
Description: The primary intervention acceptability metric will be participant ratings of overall comfort with the group program (% rating comfort with the group sessions =>4 on a single 1-5 Likert scale). Given the preliminary, open pilot nature of this protocol, the investigators will not set a priori criteria to establish acceptability but will rather use these data to inform ongoing protocol refinement.
Time Frame: Approximately 6 weeks following group program start
Measure: Count of Participants; unit: Participants
Arm/Group | Mind-Body Sexual Well-Being Group Intervention
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: Between baseline and end of program (approximately 6 weeks)
Arm/Group | Mind-Body Sexual Well-Being Group Intervention
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mind-Body Sexual Well-Being Group Intervention (N=6)
Short-term abdominal discomfort (Gastrointestinal disorders) | 2 — Determined not to be related to study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT06331403/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT06331403/ICF_001.pdf